CLINICAL TRIAL: NCT04346433
Title: Sleep and Stigma: Novel Moderators in the Relationship Between Weight Status and Cognitive Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Lindsay M Stager, Graduate Research Assistant, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: TBD2020
Record Dates: First submitted 2020-04-09; First posted 2020-04-15 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Obesity, Childhood; Overweight, Childhood
Keywords: sleep; stigma; cognitive function; nutrition
MeSH Terms: conditions — Pediatric Obesity; Social Stigma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adolescents with Normal Weight (Experimental): This group will be comprised of 30 adolescents with normal weight (BMI equal to or greater than the 5th percentile but less than the 85th percentile). Participants will be asked to engage in the sleep manipulation intervention.
  Interventions: Behavioral: Restricted Sleep; Behavioral: Adequate Sleep
- Adolescents with Overweight or Obesity (Experimental): This group will be comprised of 30 adolescents with overweight or obesity (BMI equal to or above the 85th percentile). Participants will be asked to engage in the sleep manipulation intervention.
  Interventions: Behavioral: Restricted Sleep; Behavioral: Adequate Sleep

INTERVENTIONS:
Behavioral: Restricted Sleep — During the restricted sleep condition adolescents will sleep 4 hours ±1 hour (0100-0500). This condition will last 1 night.
Behavioral: Adequate Sleep — During the adequate sleep condition adolescents will sleep 9 hours ±1 hour (2100- 0800). This condition will last 1 night.

SUMMARY:
The investigators aim to assess the relationship between overweight/obesity and decreased cognitive function in adolescents. While this relationship has been seen in past literature, the causal mechanisms are still unclear. Thus, the present study will assess sleep and stigma as possible moderators. As sleep is related to both weight and cognitive abilities it may be an important factor in the relationship between these two variables. Further, people with overweight/obesity have higher risk for stigma experiences which may increase inflammation through chronic stress and elevated cortisol. Because inflammation is theorized to play a role in the relationship between elevated BMI and decreased cognitive function, stigma may be an important moderator. 60 adolescent participants will complete two sleep conditions (adequate and restricted) in a randomized order, each followed by a lab visit during which participants will complete a short cognitive battery. At these visits, participants will also be given a self serve breakfast with a variety of whole and processed food options to further evaluate the relationship between overweight/obesity, sleep, nutritional intake, and cognitive function.

DETAILED DESCRIPTION:
Obesity represents one of our nation's leading public health issues. In 2017, over 30% of U.S. high school students had either overweight (15.6%) or obesity (14.8%), and the average U.S. BMI continues to rise. Overall, this increasing trend is associated with earlier mortality and lower quality of life. In 2005 it was projected that if current U.S. weight trends continued, the average lifespan would decrease by about 9 months. Documented declines exceed this calculation, with rises in BMI relating to an estimated 11-month decrease in life expectancy in 2011. In adolescents specifically, this epidemic shares associations with many negative health outcomes including poorer sleep quality, impaired academic performance, and lower cognitive function. Thus, it is imperative that researchers work to understand the complex nature of this preventable disease and recognize its significant longitudinal health implications.

One factor significantly related to overweight/obesity (OWOB) is decreased cognitive function. However, the causal nature of this relationship is unclear. It has been hypothesized that impaired cognitive function and poor inhibition could predict increased food consumption, thus contributing to the association between cognitive deficits and OWOB. Alternatively, it has been suggested that biological factors stemming from obesity (i.e. low grade inflammation, insulin resistance, low blood flow, and increased levels of cytokines and leptin) work to exacerbate preexisting cognitive impairments, or are perhaps fully responsible for the cognitive deficits seen in individuals with OWOB. Thus, further research is needed to clarify these relationships.

Research regarding OWOB and cognitive function has left a critical gap in the literature by failing to consider the role of sleep within this relationship. Current evidence shows that more than 2/3 of adolescents fail to attain the recommended minimum of 8 hours of sleep during the week. However, a meta-analysis found that every added hour of sleep that adolescents do secure relates to a 9.0% decrease in obesity risk. In line with this finding, sleep restriction is associated with increased appetite, hunger, and poorer nutritional food choices. Sleep restriction has also been tied to impairments in cognitive function including decreased working memory and attention. Thus, it is possible that the relationship between OWOB and cognitive function in adolescents is influenced by sleep behaviors.

Another important factor to consider in the relationship between OWOB and cognitive function is stigma. Weight stigma is a pervasive problem with multiple implications for physical health. For example, chronic low-grade inflammation represents a known correlate of chronic stress and stigmatization. This is significant as elevated inflammation also relates to OWOB and decreased cognitive function. Thus, the experience of weight related stigma may exacerbate existing inflammation in individuals with OWOB, further impairing cognitive function.

The present study seeks to expand our knowledge of these complex relationships, exploring the associations between weight status, eating behavior, cognitive function, sleep, and stigma. To do this, the study will utilize data from 2 groups: adolescents with normal weight and adolescents with OWOB. Adolescents in each group will complete two sleep conditions in a randomized order: adequate and restricted. Each sleep condition will be followed by a self-serve breakfast and completion of a cognitive battery. Prior to completing the sleep conditions, adolescents will participate in a baseline appointment during which they will complete a questionnaire regarding weight related stigma experiences.

The investigators propose that cognitive function and sleep restriction may relate to adolescent weight status through the following mechanisms: 1) elevated adiposity will predict greater impairments in cognitive functioning, poorer nutritional intake, and greater food consumption, 2) sleep restriction will result in impaired cognitive functioning, poorer nutritional intake, and increased food consumption in all adolescents, 3) sleep restriction in adolescents with elevated adiposity will result in the greatest cognitive impairments, poorest nutritional intake, and greatest food consumption, and 4) decreased cognitive function will be associated with poorer nutritional intake and greater food consumption in all adolescents. The investigators also propose that stigma experiences relate to adolescent weight status through the following mechanisms: 1) heightened stigma experiences will predict impairments in cognitive functioning in all adolescents and 2) elevated adiposity will relate to greater stigma experiences and subsequently higher cognitive impairments, resulting in the worst outcomes for assessments of cognitive function .

ELIGIBILITY:
Inclusion Criteria:

* Adolescent ages 14-19

Exclusion Criteria:

* age under 14 or over 19
* sleep disorder
* use of medications which impact sleep
* learning disorder
* history of eating disorder
* recent weight changes >10 pounds in the last 1 month
* current feeding/eating difficulties
* scores on the food fussiness sub-scale of the Childhood Eating Behaviors Questionnaire above 4.5 (out of 5)

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 61 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Objectively Measured Cognitive Function Composite Score After Sleep Restriction | Immediately after the sleep restricted intervention
  Overall cognitive function score measured using the National Institute of Health Toolbox Cognition Battery. Scores reported as standard scores with an average normative score of 100 and standard deviation of 15. Higher standard scores indicate better performance.
Objectively Measured Cognitive Function Composite Score After Adequate Sleep | Immediately after the adequate sleep intervention
  Overall cognitive function score measured using the National Institute of Health Toolbox Cognition Battery. Scores reported as standard scores with an average normative score of 100 and standard deviation of 15. Higher standard scores indicate better performance.
Objectively Measured Fluid Cognition Composite Score After Sleep Restriction | Immediately after the sleep restricted intervention
  Executive function, attention, processing speed, and episodic and working memory measured using the National Institute of Health Toolbox Cognition Battery. Scores reported as standard scores with an average normative score of 100 and standard deviation of 15. Higher standard scores indicate better performance.
Objectively Measured Fluid Cognition Composite Score After Adequate Sleep | Immediately after the adequate sleep intervention
  Executive function, attention, processing speed, and episodic and working memory measured using the National Institute of Health Toolbox Cognition Battery. Scores reported as standard scores with an average normative score of 100 and standard deviation of 15. Higher standard scores indicate better performance.
Objectively Measured Attention After Sleep Restriction | Immediately after the sleep restricted intervention
  Measured using the Flanker Inhibitory Control and Attention subtest of the National Institute of Health Toolbox Cognition Battery. Scores reported as standard scores with an average normative score of 100 and standard deviation of 15. Higher standard scores indicate better performance.
Objectively Measured Attention After Adequate Sleep | Immediately after the adequate sleep intervention
  Measured using the Flanker Inhibitory Control and Attention subtest of the National Institute of Health Toolbox Cognition Battery. Scores reported as standard scores with an average normative score of 100 and standard deviation of 15. Higher standard scores indicate better performance.
Objectively Measured Working Memory After Sleep Restriction | Immediately after the sleep restricted intervention
  Measured using the List Sorting Working Memory subtest of the National Institute of Health Toolbox Cognition Battery. Scores reported as standard scores with an average normative score of 100 and standard deviation of 15. Higher standard scores indicate better performance.
Objectively Measured Working Memory After Adequate Sleep | Immediately after the adequate sleep intervention
  Measured using the List Sorting Working Memory subtest of the National Institute of Health Toolbox Cognition Battery. Scores reported as standard scores with an average normative score of 100 and standard deviation of 15. Higher standard scores indicate better performance.
Objectively Measured Processing Speed After Sleep Restriction | Immediately after the sleep restricted intervention
  Measured using the Pattern Comparison Processing Speed subtest of the National Institute of Health Toolbox Cognition Battery. Scores reported as standard scores with an average normative score of 100 and standard deviation of 15. Higher standard scores indicate better performance.
Objectively Measured Processing Speed After Adequate Sleep | Immediately after the adequate sleep intervention
  Measured using the Pattern Comparison Processing Speed subtest of the National Institute of Health Toolbox Cognition Battery. Scores reported as standard scores with an average normative score of 100 and standard deviation of 15. Higher standard scores indicate better performance.
Objectively Measured Cognitive Flexibility After Sleep Restriction | Immediately after the sleep restricted intervention
  Measured using the Dimensional Change Card Sort subtest of the National Institute of Health Toolbox Cognition Battery. Scores reported as standard scores with an average normative score of 100 and standard deviation of 15. Higher standard scores indicate better performance.
Objectively Measured Cognitive Flexibility After Adequate Sleep | Immediately after the adequate sleep intervention
  Measured using the Dimensional Change Card Sort subtest of the National Institute of Health Toolbox Cognition Battery. Scores reported as standard scores with an average normative score of 100 and standard deviation of 15. Higher standard scores indicate better performance.
Objectively Measured Inhibition After Sleep Restriction | Immediately after the sleep restricted intervention
  Measured using the Stroop Task
Objectively Measured Inhibition After Adequate Sleep | Immediately after the adequate sleep intervention
  Measured using the Stroop Task
Objectively Measured Episodic Memory After Adequate Sleep | Immediately after the adequate sleep intervention
  Measured using the Picture Sequence Memory subtest of the National Institute of Health Toolbox Cognition Battery. Scores reported as standard scores with an average normative score of 100 and standard deviation of 15. Higher standard scores indicate better performance.
Objectively Measured Episodic Memory After Restricted Sleep | Immediately after the restricted sleep intervention
  Measured using the Picture Sequence Memory subtest of the National Institute of Health Toolbox Cognition Battery. Scores reported as standard scores with an average normative score of 100 and standard deviation of 15. Higher standard scores indicate better performance.

SECONDARY OUTCOMES:
Subjectively Measured Behavior Regulation | Baseline
  Inhibition and self-monitoring measured using the Behavior Rating Inventory of Executive Function. Scores are given as T-scores and percentiles with higher values indicating greater impairment.
Subjectively Measured Emotional Regulation | Baseline
  Emotional control and shifting measured using the Behavior Rating Inventory of Executive Function. Scores are given as T-scores and percentiles with higher values indicating greater impairment.
Subjectively Measured Cognitive Regulation | Baseline
  Task completion, working memory, and planning/organizing measured using the Behavior Rating Inventory of Executive Function. Scores are given as T-scores and percentiles with higher values indicating greater impairment.
Subjectively Measured Global Executive Composite | Baseline
  Overall score on the Behavior Rating Inventory of Executive Function. Scores are given as T-scores and percentiles with higher values indicating greater impairment.
Food Consumption After Sleep Restriction | Immediately after the sleep restricted intervention
  Participants will be given a self-serve breakfast of whole and processed foods. Foods will be weighed to the nearest 0.1g before and after the meal to determine the amount consumed. Overall macronutrient content of foods consumed will be recorded.
Food Consumption After Adequate Sleep | Immediately after the adequate sleep intervention
  Participants will be given a self-serve breakfast of whole and processed foods. Foods will be weighed to the nearest 0.1g before and after the meal to determine the amount consumed. Overall macronutrient content of foods consumed will be recorded.
Stigma Experiences | Baseline
  Measured using the brief version of the Stigmatizing Situations Inventory. Composite scores range from 0-90, with higher scores indicating more frequent stigma experiences.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron D Fobian, PhD, Study Director — The University of Alabama at Birmingham; Lindsay M Stager, Principal Investigator — The University of Alabama at Birmingham
Locations (1):
- Sparks Center, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Daniels SR, Arnett DK, Eckel RH, Gidding SS, Hayman LL, Kumanyika S, Robinson TN, Scott BJ, St Jeor S, Williams CL. Overweight in children and adolescents: pathophysiology, consequences, prevention, and treatment. Circulation. 2005 Apr 19;111(15):1999-2012. doi: 10.1161/01.CIR.0000161369.71722.10. PMID 15837955
- [Background] Liang J, Matheson BE, Kaye WH, Boutelle KN. Neurocognitive correlates of obesity and obesity-related behaviors in children and adolescents. Int J Obes (Lond). 2014 Apr;38(4):494-506. doi: 10.1038/ijo.2013.142. Epub 2013 Aug 5. PMID 23913029
- [Background] Tirosh A, Shai I, Afek A, Dubnov-Raz G, Ayalon N, Gordon B, Derazne E, Tzur D, Shamis A, Vinker S, Rudich A. Adolescent BMI trajectory and risk of diabetes versus coronary disease. N Engl J Med. 2011 Apr 7;364(14):1315-25. doi: 10.1056/NEJMoa1006992. PMID 21470009
- [Background] Lee JM, Gebremariam A, Vijan S, Gurney JG. Excess body mass index-years, a measure of degree and duration of excess weight, and risk for incident diabetes. Arch Pediatr Adolesc Med. 2012 Jan;166(1):42-8. doi: 10.1001/archpedi.166.1.42. PMID 22213749
- [Background] TODAY Study Group; Zeitler P, Hirst K, Pyle L, Linder B, Copeland K, Arslanian S, Cuttler L, Nathan DM, Tollefsen S, Wilfley D, Kaufman F. A clinical trial to maintain glycemic control in youth with type 2 diabetes. N Engl J Med. 2012 Jun 14;366(24):2247-56. doi: 10.1056/NEJMoa1109333. Epub 2012 Apr 29. PMID 22540912
- [Background] Olivo G, Gour S, Schioth HB. Low neuroticism and cognitive performance are differently associated to overweight and obesity: A cross-sectional and longitudinal UK Biobank study. Psychoneuroendocrinology. 2019 Mar;101:167-174. doi: 10.1016/j.psyneuen.2018.11.014. Epub 2018 Nov 12. PMID 30469083
- [Background] Ronan L, Alexander-Bloch A, Fletcher PC. Childhood Obesity, Cortical Structure, and Executive Function in Healthy Children. Cereb Cortex. 2020 Apr 14;30(4):2519-2528. doi: 10.1093/cercor/bhz257. PMID 31646343
- [Background] Maayan L, Hoogendoorn C, Sweat V, Convit A. Disinhibited eating in obese adolescents is associated with orbitofrontal volume reductions and executive dysfunction. Obesity (Silver Spring). 2011 Jul;19(7):1382-7. doi: 10.1038/oby.2011.15. Epub 2011 Feb 24. PMID 21350433
- [Background] Volkow ND, Wang GJ, Baler RD. Reward, dopamine and the control of food intake: implications for obesity. Trends Cogn Sci. 2011 Jan;15(1):37-46. doi: 10.1016/j.tics.2010.11.001. Epub 2010 Nov 24. PMID 21109477
- [Background] Hollmann M, Hellrung L, Pleger B, Schlogl H, Kabisch S, Stumvoll M, Villringer A, Horstmann A. Neural correlates of the volitional regulation of the desire for food. Int J Obes (Lond). 2012 May;36(5):648-55. doi: 10.1038/ijo.2011.125. Epub 2011 Jun 28. PMID 21712804
- [Background] Boeka AG, Lokken KL. Neuropsychological performance of a clinical sample of extremely obese individuals. Arch Clin Neuropsychol. 2008 Jul;23(4):467-74. doi: 10.1016/j.acn.2008.03.003. Epub 2008 Apr 29. PMID 18448310
- [Background] Galioto R, Bond D, Gunstad J, Pera V, Rathier L, Tremont G. Executive functions predict weight loss in a medically supervised weight loss programme. Obes Sci Pract. 2016 Dec;2(4):334-340. doi: 10.1002/osp4.70. Epub 2016 Sep 28. PMID 28090338
- [Background] Dassen FCM, Houben K, Allom V, Jansen A. Self-regulation and obesity: the role of executive function and delay discounting in the prediction of weight loss. J Behav Med. 2018 Dec;41(6):806-818. doi: 10.1007/s10865-018-9940-9. Epub 2018 May 25. PMID 29802535
- [Background] Butryn ML, Martinelli MK, Remmert JE, Roberts SR, Zhang F, Forman EM, Manasse SM. Executive Functioning as a Predictor of Weight Loss and Physical Activity Outcomes. Ann Behav Med. 2019 Aug 29;53(10):909-917. doi: 10.1093/abm/kaz001. PMID 30689688
- [Background] Allom V, Mullan B, Smith E, Hay P, Raman J. Breaking bad habits by improving executive function in individuals with obesity. BMC Public Health. 2018 Apr 16;18(1):505. doi: 10.1186/s12889-018-5392-y. PMID 29661241
- [Background] Alosco ML, Galioto R, Spitznagel MB, Strain G, Devlin M, Cohen R, Crosby RD, Mitchell JE, Gunstad J. Cognitive function after bariatric surgery: evidence for improvement 3 years after surgery. Am J Surg. 2014 Jun;207(6):870-6. doi: 10.1016/j.amjsurg.2013.05.018. Epub 2013 Oct 10. PMID 24119892
- [Background] Gonzales MM, Tarumi T, Miles SC, Tanaka H, Shah F, Haley AP. Insulin sensitivity as a mediator of the relationship between BMI and working memory-related brain activation. Obesity (Silver Spring). 2010 Nov;18(11):2131-7. doi: 10.1038/oby.2010.183. Epub 2010 Sep 2. PMID 20814415
- [Background] Lasselin J, Magne E, Beau C, Aubert A, Dexpert S, Carrez J, Laye S, Forestier D, Ledaguenel P, Capuron L. Low-grade inflammation is a major contributor of impaired attentional set shifting in obese subjects. Brain Behav Immun. 2016 Nov;58:63-68. doi: 10.1016/j.bbi.2016.05.013. Epub 2016 May 17. PMID 27223095
- [Background] Chen X, Beydoun MA, Wang Y. Is sleep duration associated with childhood obesity? A systematic review and meta-analysis. Obesity (Silver Spring). 2008 Feb;16(2):265-74. doi: 10.1038/oby.2007.63. No abstract available. PMID 18239632
- [Background] CDC. Sleep and sleep disorders: Data and statistics. 2017.
- [Background] Capers PL, Fobian AD, Kaiser KA, Borah R, Allison DB. A systematic review and meta-analysis of randomized controlled trials of the impact of sleep duration on adiposity and components of energy balance. Obes Rev. 2015 Sep;16(9):771-82. doi: 10.1111/obr.12296. Epub 2015 Jun 22. PMID 26098388
- [Background] Lo JC, Ong JL, Leong RL, Gooley JJ, Chee MW. Cognitive Performance, Sleepiness, and Mood in Partially Sleep Deprived Adolescents: The Need for Sleep Study. Sleep. 2016 Mar 1;39(3):687-98. doi: 10.5665/sleep.5552. PMID 26612392
- [Background] Alhola P, Polo-Kantola P. Sleep deprivation: Impact on cognitive performance. Neuropsychiatr Dis Treat. 2007;3(5):553-67. PMID 19300585
- [Background] Park H, Tsai KM, Dahl RE, Irwin MR, McCreath H, Seeman TE, Fuligni AJ. Sleep and Inflammation During Adolescence. Psychosom Med. 2016 Jul-Aug;78(6):677-85. doi: 10.1097/PSY.0000000000000340. PMID 27136501
- [Background] Dennis JA, Alazzeh A, Kumfer AM, McDonald-Thomas R, Peiris AN. The Association of Unreported Sleep Disturbances and Systemic Inflammation: Findings from the 2005-2008 NHANES. Sleep Disord. 2018 Oct 9;2018:5987064. doi: 10.1155/2018/5987064. eCollection 2018. PMID 30402295
- [Background] Beebe DW, Simon S, Summer S, Hemmer S, Strotman D, Dolan LM. Dietary intake following experimentally restricted sleep in adolescents. Sleep. 2013 Jun 1;36(6):827-34. doi: 10.5665/sleep.2704. PMID 23729925
- [Background] Wardle J, Guthrie CA, Sanderson S, Rapoport L. Development of the Children's Eating Behaviour Questionnaire. J Child Psychol Psychiatry. 2001 Oct;42(7):963-70. doi: 10.1111/1469-7610.00792. PMID 11693591
- [Background] Ancoli-Israel S, Cole R, Alessi C, Chambers M, Moorcroft W, Pollak CP. The role of actigraphy in the study of sleep and circadian rhythms. Sleep. 2003 May 1;26(3):342-92. doi: 10.1093/sleep/26.3.342. PMID 12749557
- [Background] Vartanian, L. R., Pinkus, R. T., & Smyth, J. M. (2018). Experiences of weight stigma in everyday life: Implications for health motivation. Stigma and Health, 3(2), 85-92. https://doi.org/10.1037/sah0000077
- [Background] Davis AL, Avis KT, Schwebel DC. The effects of acute sleep restriction on adolescents' pedestrian safety in a virtual environment. J Adolesc Health. 2013 Dec;53(6):785-90. doi: 10.1016/j.jadohealth.2013.07.008. Epub 2013 Sep 3. PMID 24012066
- [Background] Goldberg TE, Harvey PD, Wesnes KA, Snyder PJ, Schneider LS. Practice effects due to serial cognitive assessment: Implications for preclinical Alzheimer's disease randomized controlled trials. Alzheimers Dement (Amst). 2015 Mar 29;1(1):103-11. doi: 10.1016/j.dadm.2014.11.003. eCollection 2015 Mar. PMID 27239497
- [Background] Pilli R, Naidu M, Pingali UR, Shobha JC, Reddy AP. A computerized stroop test for the evaluation of psychotropic drugs in healthy participants. Indian J Psychol Med. 2013 Apr;35(2):180-9. doi: 10.4103/0253-7176.116251. PMID 24049230
- [Background] Sutin AR, Stephan Y, Luchetti M, Terracciano A. Perceived weight discrimination and C-reactive protein. Obesity (Silver Spring). 2014 Sep;22(9):1959-61. doi: 10.1002/oby.20789. Epub 2014 May 14. PMID 24828961
- [Background] Warren M, Beck S, Rayburn J. The State of Obesity Better Policies ofr a Healthier America. 2018.
- [Derived] Stager LM, Watson CS, Cook EW 3rd, Fobian AD. Effect of Sleep Restriction on Adolescent Cognition by Adiposity: A Randomized Crossover Trial. JAMA Neurol. 2024 Jul 1;81(7):712-721. doi: 10.1001/jamaneurol.2024.1332. PMID 38767872